CLINICAL TRIAL: NCT04135924
Title: Influence of Trainning Respiratory Muscle About Gate and Physiological and Functional Variables in Parkinson's Disease
Brief Title: Influence of Trainning in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Metodista de Piracicaba (Other)
Collaborators: Universidade do Estado do Pará (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, Director of Human Movement Department, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 031.819.852-52
Record Dates: First submitted 2019-03-28; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease
Keywords: Rehabilitation; Neurological disease
MeSH Terms: conditions — Parkinson Disease; Nervous System Diseases | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- walking nordic and respiratory training group (Active Comparator): It will be composed of patients with clinical diagnosis of Parkinson's disease, who will be submitted to respiratory muscle training (TMR) associated with the Nordic walking(NC) training .
  Interventions: Other: Rehabilitation
- walking nordic group (Active Comparator): It will be composed of patients with clinical diagnosis of Parkinson's disease, who will only be submitted to Nordic walking training.
  Interventions: Other: Rehabilitation
- respiratory training group (Active Comparator): It will be composed of patients with clinical diagnosis of Parkinson's disease, who will only be submitted to respiratory muscle training protocol.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — physical exercise and respiratory muscle training

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disorder of the central nervous system (CNS), chronic and progressive that is associated with the loss of dopaminergic neurons in the compact part of the substantia nigra.

These patients often show excessive fatigue and dyspnea with the progression of the disease, and the later onset of treatment, lower the tolerance of the patient to perform physical activities.

Walking is one of the main limiting factors for a good quality of life. Therefore, gait training can promote individuals a better physical condition to recover their activities, as well as to maintain good posture, and reduce exacerbated flexion of the characteristic spine, preventing falls and various types of trauma. A proposed gait training is the Nordic walk, which, when using sticks to gain balance, stability and coordination, allows the individual to obtain better functional capacity, besides performing aerobic and stimulating activity.

In addition to the gait training, this research proposes respiratory muscle training (TMR), using a linear resistor capable of promoting resistance and strength gain of the inspiratory musculature. TMR is a therapeutic modality consecrated in the maximal inspiratory and expiratory pressure gain, directly influencing the peripheral musculature, favoring the practice of physical activities, such as walking itself to possibly condition the patient to longevity and dignity to practice their ADLs with better quality of life, allowing delayed disease progression.

In addition, the practice of these individuals submitted to walking and respiratory muscle training protocols can bring great benefits as regards their quality of life, and their perception of space, as well as their importance in the social environment. One form of evidence to qualify these aspects is the quality of life assessment scale in PDQ-39 Parkinson's Disease Patients, which contributes among other factors to the satisfaction and performance of the activity.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder of the central nervous system (CNS), chronic and progressive that is associated with the loss of dopaminergic neurons in the compact part of the substantia nigra ( AYANO , 2016). Its clinical diagnosis is due to a set of signs and symptoms, initially observed for the motor characteristics that may be: rest tremor, bradykinesia, postural instability, festinating gait and joint stiffness, which directly interfere in the quality of life of these individuals ( CUGUSI and t al., 2017).

Some studies have shown that patients with PD exhibit multiple respiratory symptoms , including reduced respiratory muscle strength, rapid and coordinated action performance impairment, efficient contractions of the chest wall musculature, and effective cough reduction. With the progression of the disease, these limitations can trigger aspiration pneumonia, which is the main cause of death in this profile of individuals ( TROCHE et al ., 2010 ; SAPIENZA et al., 2011; JÚNIOR et al., 2015 ).

From the epidemiological point of view, feta accounts for about 1% of the population over 65 years and more than 3% after 75 years of age, with an incidence of 1.5 men over women. ( SILVA, 2018). The projection for 2030 is that more than 8 million individuals over the age of 60 have Parkinson's disease. In the United States about 59,000 new cases emerge every year. In Brazil, epidemiological data on the disease are still scarce, but it is estimated that around 200,000 people have the disease ( FERNANDES; FILHO, 2018 ).

These patients often show excessive fatigue and dyspnea with the progression of the disease, and the later onset of treatment, lower the tolerance of the patient to perform physical activities.Therefore, it is sought through health promotion to guide the need for physical practice through exercises that can contribute to the improvement of their quality of life and in the previous training of the respiratory muscles, influencing the main functional skills, such as am archa. ( REYES, CASTILLO et al., 2018; RASSLER et al., 2011).

Walking is one of the main limiting factors for a good quality of life. Therefore, gait training can promote individuals a better physical condition to recover their activities, as well as to maintain good posture, and reduce exacerbated flexion of the characteristic spine, preventing falls and various types of trauma. A proposed gait training is the Nordic walk, which, when using sticks to gain balance, stability and coordination, allows the individual to obtain better functional capacity, besides performing aerobic and stimulating activity (XU et al., 2018) .

In addition to the gait training, this research proposes respiratory muscle training (TMR), using a linear resistor capable of promoting resistance and strength gain of the inspiratory musculature. TMR is a therapeutic modality consecrated in the maximal inspiratory and expiratory pressure gain, directly influencing the peripheral musculature, favoring the practice of physical activities, such as walking itself to possibly condition the patient to longevity and dignity to practice their ADLs with better quality of life, allowing delayed disease progression (Júnior et al., 2015).

In addition, the practice of these individuals submitted to walking and respiratory muscle training protocols can bring great benefits as regards their quality of life, and their perception of space, as well as their importance in the social environment. One form of evidence to qualify these aspects is the quality of life assessment scale in PDQ-39 Parkinson's Disease Patients, which contributes among other factors to the satisfaction and performance of the activity (JA et al., 2012; ).

Thus, the objective of this study is to verify the influence of respiratory muscle training associated with Nordic walking training on the physiological, biochemical and functional variables in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* without cognitive impairment
* Mini Mental State Examination with scores above 23
* clinical diagnosis of Parkinson's disease in grade 2-3 on the scale modified Hoehn and Yarh

Exclusion Criteria:

* volunteers who present cognitive, auditory and visual alterations, that incapacitate them to carry out the proposed procedure
* carriers of Diabetes Mellitus and other metabolic diseases
* heart disease and uncontrolled hypertension
* ethyl alcohol
* smoker
* those hospitalized at least six months prior to the study
* as well as those who do not use the medication and the correct dosage prescribed by the physician
* individuals with osteomioarticular dysfunctions and neurological diseases
* restricted to wheelchairs

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of lipid peroxidation | 8 weeks
  Oxigen-reactive species
Respiratory function | 8 weeks
  spirometry variables analysis

CONTACTS AND LOCATIONS:
Overall Officials: Lucas M Matos, graduated, Study Chair — Universidade do Estado do Pará
Locations (1):
- Universidade do Estado do Pará, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Earhart GM, Falvo MJ. Parkinson disease and exercise. Compr Physiol. 2013 Apr;3(2):833-48. doi: 10.1002/cphy.c100047. PMID 23720332
- [Result] Hoehn MM, Yahr MD. Parkinsonism: onset, progression, and mortality. 1967. Neurology. 2001 Nov;57(10 Suppl 3):S11-26. No abstract available. PMID 11775596
- [Result] Reyes A, Castillo A, Castillo J, Cornejo I. The effects of respiratory muscle training on peak cough flow in patients with Parkinson's disease: a randomized controlled study. Clin Rehabil. 2018 Oct;32(10):1317-1327. doi: 10.1177/0269215518774832. Epub 2018 May 13. PMID 29756459
- [Result] Reyes A, Ziman M, Nosaka K. Respiratory muscle training for respiratory deficits in neurodegenerative disorders: a systematic review. Chest. 2013 May;143(5):1386-1394. doi: 10.1378/chest.12-1442. PMID 23714850
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886